CLINICAL TRIAL: NCT03668457
Title: Effectiveness and Cost-effectiveness of a Multi-component Intervention to Improve Medication Adherence in People With Depressive Disorders
Brief Title: A Multi-component Intervention to Improve Medication Adherence in People With Depressive Disorders
Acronym: MAPDep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Servicio Canario de Salud (Other)
Collaborators: University of La Laguna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: PI18-00767
Record Dates: First submitted 2018-07-09; First posted 2018-09-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Depressive Disorder
Keywords: Depression; Medication adherence; Multicomponent intervention
MeSH Terms: conditions — Depressive Disorder; Depression; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention to Patients (Experimental): Only patients receive intervention
  Interventions: Behavioral: Intervention to Patients; Other: Control
- Intervention to Psychiatrists (Experimental): Psychiatrists receive the intervention. Their associated patients do not receive direct intervention although indirect intervention through professionals
  Interventions: Behavioral: Intervention to Psychiatrists; Other: Control
- Mixed Intervention (Experimental): Patients and Psychiatrists associated with these patients receive intervention
  Interventions: Behavioral: Intervention to Patients; Behavioral: Intervention to Psychiatrists; Other: Control
- Control (Other): Psychiatrists provide the usual care Patients receive usual care
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Intervention to Patients — Multifaceted intervention consisting of:
  1. A collaborative care management intervention, including depression education, medication management and behavioral activation.
  2. Use of a medication reminder mobile app.
  Arms: Intervention to Patients; Mixed Intervention
Behavioral: Intervention to Psychiatrists — Educational intervention consisting of theoretical and practical sessions to to improve communication and negotiation abilities, and to develop skills to promote patient-centered care and shared decision-making.
  Arms: Intervention to Psychiatrists; Mixed Intervention
Other: Control — Other: Usual care Usual care for depressive disorder received in mental health units

SUMMARY:
Objective: The study of medication adherence in depression (MAPDep study) aims to evaluate the effectiveness and cost-effectiveness of a multi-component strategy to enhance patient-centered care to improve adherence toward medications in patients with depression, formed by an educational intervention to psychiatrists and/or a collaborative care intervention group to patients and relatives plus a reminder system through the use of a mobile APP.

Methods: The objective will be assessed under an open multicenter, clinical controlled trial with random allocation by clusters to one of three interventions or to usual care (control arm). In group 1 only patients and family members receive intervention, in group 2 only psychiatrists receive intervention, and group 3 is a combined intervention for patients and psychiatrists. The main measure will be the change in medication adherence rate. Secondary endpoints are depression, emotional distress, health-related quality of life, physical functioning, patients' knowledge about their medications, provider beliefs regarding patient-centeredness, and healthcare resource utilization.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  * Patients with diagnosis of depressive disorder (major depressive disorder MDD and/or dysthymia) under pharmacological treatment
  * Regular users of mobile phones
  * Patients who have consulted their psychiatrist about their depression at least once in the previous 6 months
* Health professionals:

Psychiatrists have no intention of moving from their practice during the study period.

Exclusion criteria:

• Patient:

* Patients with history of current bipolar disorder and/or any psychotic disorder
* Insufficient language skills
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Change in the Sidorkiewicz instrument score | Baseline and 6 months
  Change in adherence from baseline to 6 months. This instrument contains 5 questions to help patients recognize their different medication-taking behaviors for each drug taken. The results generate adherence levels ranging from 1 (high drug adherence) to 6 (drug discontinuation).

SECONDARY OUTCOMES:
Change in the Sidorkiewicz instrument score | Baseline, 3 and 12 months
  Change in adherence from baseline to 3 and 12 months.
Change in Beck Depression Inventory - II (BDI-II) score | Baseline, 3, 6, and 12 months
  BDI-II contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms.
Change in Hospital Anxiety and Depression Scale (HADS) score | Baseline, 3, 6, and 12 months
  HADS contains two 7-item Likert scales, one for anxiety and one for depression, with responses being scored on a scale of 0-3 (3 indicates higher symptom frequencies).
Change in Physical Functioning Subscale (PF-10) of the 36-item Short Form Health Survey (SF-36) | Baseline, 6, and 12 months
  PF-10 contains 10-item Likert scale designed to examine a person's perceived limitation with physical functioning. Each item is rated on a 3-point scale (yes, limited a lot; yes, limited a little; and no, not limited at all).
Change in EQ-5D-5L | Baseline, 6, and 12 months
  EQ-5D-5L is a questionnaire consisting of five domains (Mobility, Self-Care, Usual Activity, Pain/Discomfort and Anxiety/Depression) each with five levels (no problems, slight problems, moderate problems, severe problems and extreme problems).
Change in Patient-Practitioner Orientation Scale (PPOS) score | Baseline and 12 months
  PPOS is a self-administered questionnaire that assesses patient-centeredness healthcare professionals. PPOS contains 18 items scored on a 6-point Likert scale (strongly disagree to strongly agree).

OTHER OUTCOMES:
Healthcare utilization, cost and productivity losses | Baseline, 6, and 12 months
  Costs because of the clinical management in all groups will be assessed from the healthcare services perspective, including the costs related to the development and use of all components for each intervention assessed (group sessions, app, etc.). Information about prescribed medication and doses; patient contacts with psychiatric and primary care services; hospital admissions and length of stay; and productivity losses will be obtained from a self-administered questionnaire.
The Control Preferences Scale (CPS) | Baseline
  CPS consists of five "cards" on a board, each illustrating a different role in decision-making by means of a cartoon and short descriptive statement. Patients has to choose between the cards, observing them one at a time, to establish an order of preference that ranged from a completely active role to a more passive style (from 0 to 5, where the higher the score, the more passive the style).
Drug Attitude Inventory (DAI) | Baseline
  DAI is 10-item self-report scale that assesses psychiatric patients' attitudes toward their psychopharmacological medications. Response options are true/false, with scores ranging from a minimum of -10 to a maximum of 10. A positive total score means a positive attitude, while a negative total score indicates a negative attitude.
Form C of the Multidimensional Health Locus of Control Scales (MHLC-C) | Baseline
  MHLC-C is an 18-item self-report scale composed of four subscales that measure control variables with regard to participants' health, with a 6-point rating scale ranging from 1 (strongly disagree) to 6 (strongly agree). Higher scores on each subscale indicate a stronger belief in that kind of control.
The Hong Psychological Reactance Scale (HPRS) | Baseline
  HPRS is a 14-item self-report questionnaire designed to measure the individual difference in reactance proneness. Each item is rated on a five-point Likert scale (ranging from 1 = strongly disagree to 5 = strongly agree).
Beliefs about Medicines Questionnaire (BMQ) | Baseline
  BMQ assesses patients' beliefs and worries about taking medication for their disease. It comprises a general and a specific scale.The BMQ-General scale assesses more general beliefs or social representations of pharmaceuticals as a class of treatment and includes eight items in two subscales (four items each), Overuse and Harm. The BMQ-Specific scale assesses patient's beliefs about the medication he/she is prescribed for a specific illness in terms of the necessity and concern about taking it. This scale includes ten items in two subscales (five items each), Concern and Necessity. The degree of agreement with each statement is indicated on a five-point Likert scale (ranging from 1=strongly disagree to 5=strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: María del Mar Trujillo Martín, PhD, Principal Investigator — Servicio de Evaluación del Servicio Canario de la Salud; Carlos de las Cuevas Castresana, MD, PhD, Principal Investigator — University of La Laguna; Tasmania del Pino-Sedeño, PhD, Principal Investigator — University of La Laguna
Locations (1):
- Servicio de Evaluación. Servicio Canario de Salud, Santa Cruz de Tenerife, Spain

REFERENCES:
- [Derived] Del Pino-Sedeno T, Penate W, de Las Cuevas C, Valcarcel-Nazco C, Fumero A, Serrano-Perez PG, Acosta Artiles FJ, Ramos Garcia V, Leon Salas B, Bejarano-Quisoboni D, Trujillo-Martin MM. Effectiveness and cost-effectiveness of a multicomponent intervention to improve medication adherence in people with depressive disorders - MAPDep: a study protocol for a cluster randomized controlled trial. Patient Prefer Adherence. 2019 Feb 22;13:309-319. doi: 10.2147/PPA.S172963. eCollection 2019. PMID 30863020